CLINICAL TRIAL: NCT06333522
Title: Losartan Use to Mitigate Arthrofibrosis Following Total Joint Arthroplasty
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study team unable to identify method for approval of the medication as standard of care and compounded.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-00979
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Arthrofibrosis of Knee
Keywords: Total Knee Arthroplasty (TKA)
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Losartan cohort (Experimental): Patients will initiate Losartan treatment 2 weeks pre-operatively and will continue until 4 weeks post-operatively. Range of motion will be measured as part of standard of care at the time of enrollment and at post-op office visits 2-4 weeks, 4-8 weeks and 8-20 weeks post-operatively.
  Interventions: Drug: Losartan
- Control cohort (No Intervention): No additional steps in management are required for the control arm of the study. Range of motion will be measured as part of standard of care at the time of enrollment and at post-op office visits 2-4 weeks, 4-8 weeks and 8-20 weeks post-operatively.

INTERVENTIONS:
Drug: Losartan — Patients will receive Losartan 12.5mg orally twice daily beginning 2 weeks preoperatively and continuing for 4 weeks postoperatively.
  Arms: Losartan cohort

SUMMARY:
The purpose of this study is to determine the effect of Losartan, an Angiotensin II Receptor Blocker (ARB), on the formation development of arthrofibrosis in patients who have had a primary total knee arthroplasty. This study aims to assess the post-operative range of motion and the incidence of MUA within three months following the index arthroplasty in the treatment arm (losartan) and the control arm.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are candidates for elective primary total knee arthroplasty for a diagnosis of osteoarthritis or inflammatory arthritis.
2. Patients ≥18 years of age
3. Patients have been medically cleared and scheduled for surgery
4. Patients' primary care physician has verified that the patient can safely take the described dose of Losartan for the duration of the study period.

Exclusion Criteria:

1. Patients already taking Losartan will not be included in the prospective study
2. Patients already taking an ARB (angiotensin receptor blockers) or other ACE (Angiotensin-converting-enzyme) inhibitor
3. Low blood pressure
4. Currently taking hypertensive medication
5. Revision surgery
6. Surgery for fracture, infection, or malignancy
7. Patients with a diagnosis of post-traumatic arthritis
8. Bilateral, simultaneous surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in range of motion | Baseline, Day 90
Rate of manipulation under anesthesia (MUA) after elective total knee arthroplasty | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Rozell, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Joshua.Rozell@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Joshua.Rozell@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.